CLINICAL TRIAL: NCT05999955
Title: An Open-label, Randomized, Active-controlled Study to Evaluate the Safety of Postbiotic Nasal Spray Using Inactivated DSM32444 Spores in the Treatment of Acute Rhinosinusitis, as Compared With Neomycin/ Dexamethasone/Xylometazoline Spray
Brief Title: Safety and Efficacy of DSM 32444 Postbiotic in the Treatment of Acute Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huro Biotech Joint Stock Company (Industry)
Collaborators: Vietstar Biomedical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSP32444.02
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Rhinosinusitis; Rhinitis
Keywords: Acute Rhinosinusitis; Chronic Rhinosinusitis; Allergic Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis; Rhinitis; Rhinitis, Allergic, Perennial | interventions — Neomycin; xylometazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Subjects in Control group receive Neomycin Nasal Spray for 10 days.
  Interventions: Drug: Neomycin/ Dexameythasone/Xylometazoline
- SPEROVID (Experimental): Subjects in Experimental group receive a nasal spray containing Bacillus subtilis DSM32444 ("Sperovid") for 10 days.
  Interventions: Combination Product: Bacillus subtilis DSM32444

INTERVENTIONS:
Drug: Neomycin/ Dexameythasone/Xylometazoline — The active-control in the phase II study was a commercial form of nasal spray containing Dexamethasone/Neomycin/Xylometazoline. This formulation is approved by Vietnam's Ministry of Health as a treatment regime for rhinosinusitis. Dexamethasone sodium phosphate is fluoromethyl prednisolone, a synthetic glucocorticoid. Dexamethasone has the main effects of glucocorticoids as anti-inflammatory, antiallergic and immunosuppressant. Neomycin sulfate is an antibiotic belonging to the group of aminoglycosides that have a bactericidal mechanism due to inhibition of bacterial protein biosynthesis. In this study, the nasal spray is used as an adjunct to Amoxicillin/Clavulanate standard treatment
  Arms: Control
Combination Product: Bacillus subtilis DSM32444 — Postbiotic DSM32444 is manufactured by HURO BIOTECH Company as a drug-grade active pharmaceutical ingredient. The Class A medical device containing Postbiotic DSM32444 is called Sperovid, which is manufactured by Dong Duoc Viet under ISO 13485:2016 standards for medical device. Sperovid has registration number: 220000033/ PCBALA In this study, the nasal spray is used as an adjunct to Amoxicillin/Clavulanate standard treatmen.
  Other Names: Sperovid, Speromed, Sperokid, inactivated DSM32444
  Arms: SPEROVID

SUMMARY:
Rhinitis is a type of upper respiratory infection with a common nasal pathology especially in Southeast Asia, which is characterized by the presence of one or more of the following symptoms: itchy nose, sneezing, runny nose, and nasal congestion. Other symptoms occasionally experienced include headache, excessive pain reaction, cough, fever. Rhinitis can be idiopathic or due to a variety of causes, including allergens, medications, endocrine/metabolic, infectious, inflammatory, and abnormal nasal structures. The treatment of acute rhinosinusitis and allergic rhinitis in hospitals is currently carried out according to the general professional guidance of the Vietnam Ministry of Health. Most patients are prescribed corticosteroids, antihistamines, and antibiotics for immediate decongestion and anti-inflammatory effects. Current concerns about antimicrobial resistance (AMR) as well as side effects of corticosteroids and antihistamines have led to an urgent need for a naturebased next generation therapeutic approach that is safe, effective and helps in addressing the issues of AMR. The goal of this interventional study is to evaluate the safety and efficacy of postbiotic nasal spray using inert bioparticles of Bacillus subtilis DSM32444 in treatment of acute rhinosinusitis; and to compare the efficacy against Neomycin/Dexamethasone//Xylometazoline administered as a nasal spray as an adjunct to Amoxicillin/Clavulanate standard treatment in patients with acute rhinosinusitis.

Patients with acute rhinosinusitis who give consent to participate in the study will be randomly assigned in a 1:1 ratio to one of two groups using postbiotic of Bacillus subtilis DSM32444 nasal spray ("Sperovid") or Neomycin/ Dexamethasone nasal spray for a period of 10 days. Investigators will compare whether the nasal spray using postbiotic Bacillus subtilis DSM32444 has similar efficacy as compared to Neomycin/Dexamethasone/Xylometazoline nasal spray as an adjuvant therapy along with the standard Amoxicillin/Clavulanate regimen in patients with acute rhinosinusitis based on time to improvement of rhinosinusitis symptoms.

DETAILED DESCRIPTION:
Rhinitis is a type of upper respiratory infection with a common nasal pathology especially in Southeast Asia, which is characterized by the presence of one or more of the following symptoms: itchy nose, sneezing, runny nose, and nasal congestion. Other symptoms occasionally experienced include headache, excessive pain reaction, cough, fever. Rhinitis can be idiopathic or due to a variety of causes, including allergens, medications, endocrine/metabolic, infectious, inflammatory, and abnormal nasal structures. Rhinosinusitis in general is not a dangerous pathological condition, however the frequency of the disease is relatively high with statistics showing that all people experience it at least once in their lives. Common rhinosinusitis symptoms include severe facial pains and difficulties in breathing. Hence, most patients are prescribed corticosteroids, antihistamines, and antibiotics for immediate decongestion and anti-inflammatory effects. A common treatment regime for patients with rhinosinusitis in Vietnam includes a combination of steroids and antibiotics (Neomycin/Dexamethasone/Xylometazoline) administered as a nasal spray, in adjunct with Amoxicillin/clavulanate 875/125 mg taken orally every 12 hours. Dexamethasone sodium phosphate is fluoromethyl prednisolone, a synthetic glucocorticoid. Glucocorticoids work by binding to receptors in cells, translocating into the cell nucleus, and there, affecting certain translated genes.

Glucocorticoids also have some direct effects, possibly through receptormediated attachment. Dexamethasone has the main effects of glucocorticoids as anti-inflammatory, antiallergic and immunosuppressant. In terms of anti-inflammatory activity, dexamethasone is 30 times stronger than hydrocortisone, 7 times stronger than prednisone. Neomycin sulfate is an antibiotic belonging to the group of aminoglycosides that have a bactericidal mechanism due to inhibition of bacterial protein biosynthesis. Bacteria sensitive to neomycin include: Staphylococcus aureus, Escherichia coli, Haemophilus influenzae, Klebsiella, Enterobacter of all kinds, Neisseria of all kinds. The antibiotic is used to prevent bacterial infection and is formulated for use together with glucocorticoids for a fast relief of rhinosinusitis symptoms. The duration of treatment for patients is about 10 days depending on the severity of the disease. During the treatment period, a change in the systemic antibiotic regimen is necessary if the observations after 3 to 5 days of treatment do not show signs of a satisfactory response. Current concerns about antimicrobial resistance (AMR) as well as the documented side effects of corticosteroid and antihistamine have led to an urgent need for a nature-based next generation therapeutic approach that is safe, effective and helps in addressing the AMR problem. Preclinical studies of inactivated Bacillus subtilis strain DSM32444 conducted by collaborating UK universities and laboratories have shown potential therapeutic benefits with anti-inflammatory mechanisms that may be useful in other viral infections of the respiratory tract. The reason for using an inactivated spore is because various publications have identified risks of inhalation of high doses of live bacteria in the respiratory tract and lungs. DSM32444 also carries GRAS status for human use. An accredited, cGLP, repeat-dose toxicology study also confirmed complete safety in rodent models after high doses of treatment. The investigators think there is a likelihood to apply this postbiotic technology to mitigate the overuse of antibiotics, corticosteroids, and antihistamines. The aim of this study is to evaluate the safety of a nasal spray using a postbiotic preparation of Bacillus subtilis DSM32444 and that is a sterile inert bioparticle, as well as the efficacy in treating acute rhinosinusitis as compared to Neomycin/ Dexamethasone/ Xylometazoline administered as a nasal spray.

* Study population: Sample size is 60 volunteered patients with acute rhinosinusitis.
* Description of Sites: the study is carried out at Thai Binh University of Medicine and Pharmacy and Thai Binh University of Medicine and Pharmacy Hospital.
* Description of Study intervention:

This phase is a randomized, parallel controlled, open-label, product-controlled study (Neomycin/Dexamethasone/Xylometazoline nasal spray). The randomization is carried out according to the 4-block strategy using envelopes with predetermined random codes. Study subjects will be given codes in turn sealed in sequentially numbered envelopes. The research product is formulated as an open label due to the different shape of the product. Participants in the study who are patients with rhinosinusitis (viral, bacterial or suspected bacterial) are randomly assigned in a 1:1 ratio to one of two groups using Sperovid or Neomycin/Dexamethasone/Xylometazoline nasal spray for a period of 10 days. The research product (Sperovid or Neomycin/Dexamethasone/Xylometazoline nasal spray) is sprayed 2-3 times daily, sprayed on both sides of the nose, each time 1-2 sprays corresponding to 0.2 ml/spray. Both groups of patients received amoxicillin/clavulanate 875/125 mg orally every 12 hours a day with a 10-day course of treatment. Daily nasopharyngeal symptom assessment (TSS) is performed using a diary from Day 1 to Day 10 (end of regime). The response assessment is done on Day 5 (±1) and the decision to continue or change the treatment regimen will be made by the research physician at this time.

* The study data after collection will be analyzed statistically using SAS 9.4. The normal distribution of statistical samples will be evaluated by the Kolmogorov-Smirnov-Lilliefors test, the uniformity of variance will be verified by Levene's test. The continuous variables will be analyzed using a two-dimensional variance test or covariance analysis (ANOVA/ANCOVA) in the case of a normal distribution and using the ANOVA non-parametric Kruskal-Wallis test in the case of a non-standard distribution. Repeatable measurement analyses will be used where appropriate. Differences between treatment groups in terms of duration of major symptoms of acute respiratory infection and average time to resolution will be assessed using the Student's t-test or the Mann-Whitney test. Chi-Square (or Fisher's exact test) will be used to evaluate the difference between the ratios. Analysis of classification data is carried out using the Cochran-Mantel- Haenszel test. In the absence of further note, the continuous variables are expressed by the mean ± standard deviation. The Cox analysis model and log-rank testing will be used to compare variables of the time type leading up to an event.
* Expected outcomes: (1) The nasal spray using a postbiotic preparation of Bacillus subtilis DSM32444 and that is a sterile inert bioparticle ("Sperovid") is safe and well tolerated among healthy volunteers, and (2) The inactivated Bacillus subtilis DSM32444 ("Sperovid") has similar efficacy as compared to Neomycin/Dexamethasone as an adjuvant therapy along with the standard Amoxicillin/Clavulanate regimen in patients with acute rhinosinusitis based on time to improvement of rhinosinusitis symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed rhinosinusitis patients (according to Vietnam's MOH guidelines for diagnosis of rhinosinusitis), ≥18 years of age, at the time of signing the informed consent.
* Must be in generally good health, except rhinosinusitis
* Patients who are able to use an e-Diary or Paper Diary during the study to report their health status
* Patients capable of giving a signed informed consent form (ICF)

Exclusion Criteria:

* Presence of any nasal mucosal erosion, nasal ulceration, or nasal septal perforation (Grade 1b - 4)
* Other nasal disease(s) likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa, clinically significant polyposis, or nasal structural abnormalities.
* Nasal surgery or sinus surgery within the previous year
* Chronic sinusitis - more than 3 episodes per year
* Asthma (with the exception of mild, intermittent asthma). Subjects with mild, intermittent asthma who only require short-acting inhaled bronchodilators (not more often than twice per week) and who do not have nocturnal awakening as a result of asthma are eligible for enrolment.
* Planned travel outside of the study area during the study period.
* Use of any investigational drug within 30 days prior to Day screening. No investigational products are permitted for use during the conduct of this study.
* Existence of any medical condition, which in the opinion of the investigator, might significantly affect the subject's ability to complete this trial; or their safety in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
To compare efficacy following multiple doses of the SPEROVID Nasal Spray for 10 days with those of the Neomycin/ Dexamethasone/Xylometazoline Nasal Spray in Acute Rhinosinusitis Patients assessed by time to symptom resolution | Day 1 to Day 10
  Time to symptom resolution based on total symptom score (TSS)
  TSS includes the following symptoms, each will be scored from 0 to 6:
  * Nasal obstruction/blockage/congestion
  * Discoloured nasal drainage: anterior/posterior
  * Headache
  * Fatigue
  * Decreased sense of smell
  * Ear pain/pressure/fullness
  * Cough
  * Halitosis
  * Dental pain
  * Fever
  Score Descriptions 0 or 1 None - to an occasional limited episode 2 or 3 Mild - Steady symptoms but easily tolerable 4 or 5 Moderately bothersome - Symptoms hard to tolerate, might interfere with activities of daily living, sleep, or both 6 Very severe - Symptoms are so bad that person cannot function virtually all the time

SECONDARY OUTCOMES:
To compare safety following multiple doses of the SPEROVID Nasal Spray for 10 days with those of the Neomycin/ Dexamethasone/Xylometazoline Nasal Spray in Influenza Patients | Day 1 to Day 10
  * Incidence of Adverse Events (Nasal Congestion, Itchy Nose, Allergic Reaction/Rash, Sneezing, Nasal Discharge, Weeping, Itchy eyes, Itchy ears, Sore throat, Nausea/Vomiting)
  * Incidence of Serious Adverse Events (Adverse events leading to discontinuation of study products, Adverse events leading to withdrawal of subjects from the study, Deaths up to the time of study data cut off)
  * Incidence of Related Adverse Events
  * Incidence of Related Serious Adverse Events
To compare the efficacy following multiple doses of SPEROVID Nasal Spray for 10 days with those of Neomycin/ Dexamethasone/Xylometazoline Nasal Spray in Acute Rhinosinusitis Patients assessed by time to symptom improvement | Day 1 to Day 10
  Time to symptom significant improvement based on total symptom score (TSS)
  TSS is defined in the description of Primary Outcome
To compare the efficacy following multiple doses of the SPEROVID Nasal Spray for 10 days with those of the Neomycin/Dexamethasone/Xylometazoline Nasal Spray in Acute Rhinosinusitis Patients assessed by Change From Baseline in Total Symptom Score (TSS) | Day 1 to Day 10
  Change From Baseline in Total Symptom Score (TSS)
  TSS is defined in the description of Primary Outcome
To compare the efficacy following multiple doses of the SPEROVID Nasal Spray for 10 days with those of the Neomycin/Dexamethasone/Xylometazoline Nasal Spray in Acute Rhinosinusitis Patients assessed by Clinical Failure Rate at the End of Treatment | Day 1 to Day 10
  Clinical failure is defined as the persistence of 1 or more signs and symptoms of rhinosinusitis or patients who have received additional (or new) antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Kien T NGUYEN, PhD, Principal Investigator — Thai Binh University of Medicine and Pharmacy
Locations (1):
- Thai Binh University of Medicine and Pharmacy, Thái Bình, Thai Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James J, Meyer SM, Hong HA, Dang C, Linh HTY, Ferreira W, Katsande PM, Vo L, Hynes D, Love W, Banyard AC, Cutting SM. Intranasal Treatment of Ferrets with Inert Bacterial Spores Reduces Disease Caused by a Challenging H7N9 Avian Influenza Virus. Vaccines (Basel). 2022 Sep 19;10(9):1559. doi: 10.3390/vaccines10091559. PMID 36146637
- [Background] de Souza RD, Batista MT, Luiz WB, Cavalcante RC, Amorim JH, Bizerra RS, Martins EG, Ferreira LC. Bacillus subtilis spores as vaccine adjuvants: further insights into the mechanisms of action. PLoS One. 2014 Jan 27;9(1):e87454. doi: 10.1371/journal.pone.0087454. eCollection 2014. PMID 24475289
- [Background] Huang JM, La Ragione RM, Nunez A, Cutting SM. Immunostimulatory activity of Bacillus spores. FEMS Immunol Med Microbiol. 2008 Jul;53(2):195-203. doi: 10.1111/j.1574-695X.2008.00415.x. Epub 2008 Apr 21. PMID 18430003
- [Background] Wallace DV, Dykewicz MS, Bernstein DI, Blessing-Moore J, Cox L, Khan DA, Lang DM, Nicklas RA, Oppenheimer J, Portnoy JM, Randolph CC, Schuller D, Spector SL, Tilles SA; Joint Task Force on Practice; American Academy of Allergy; Asthma & Immunology; American College of Allergy; Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. The diagnosis and management of rhinitis: an updated practice parameter. J Allergy Clin Immunol. 2008 Aug;122(2 Suppl):S1-84. doi: 10.1016/j.jaci.2008.06.003. No abstract available. PMID 18662584
- [Background] Baraniuk JN. Pathogenic mechanisms of idiopathic nonallergic rhinitis. World Allergy Organ J. 2009 Jun 15;2(6):106-14. doi: 10.1097/WOX.0b013e3181aadb16. PMID 24229057
- [Background] Bousquet J, Khaltaev N, Cruz AA, Denburg J, Fokkens WJ, Togias A, Zuberbier T, Baena-Cagnani CE, Canonica GW, van Weel C, Agache I, Ait-Khaled N, Bachert C, Blaiss MS, Bonini S, Boulet LP, Bousquet PJ, Camargos P, Carlsen KH, Chen Y, Custovic A, Dahl R, Demoly P, Douagui H, Durham SR, van Wijk RG, Kalayci O, Kaliner MA, Kim YY, Kowalski ML, Kuna P, Le LT, Lemiere C, Li J, Lockey RF, Mavale-Manuel S, Meltzer EO, Mohammad Y, Mullol J, Naclerio R, O'Hehir RE, Ohta K, Ouedraogo S, Palkonen S, Papadopoulos N, Passalacqua G, Pawankar R, Popov TA, Rabe KF, Rosado-Pinto J, Scadding GK, Simons FE, Toskala E, Valovirta E, van Cauwenberge P, Wang DY, Wickman M, Yawn BP, Yorgancioglu A, Yusuf OM, Zar H, Annesi-Maesano I, Bateman ED, Ben Kheder A, Boakye DA, Bouchard J, Burney P, Busse WW, Chan-Yeung M, Chavannes NH, Chuchalin A, Dolen WK, Emuzyte R, Grouse L, Humbert M, Jackson C, Johnston SL, Keith PK, Kemp JP, Klossek JM, Larenas-Linnemann D, Lipworth B, Malo JL, Marshall GD, Naspitz C, Nekam K, Niggemann B, Nizankowska-Mogilnicka E, Okamoto Y, Orru MP, Potter P, Price D, Stoloff SW, Vandenplas O, Viegi G, Williams D; World Health Organization; GA(2)LEN; AllerGen. Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 update (in collaboration with the World Health Organization, GA(2)LEN and AllerGen). Allergy. 2008 Apr;63 Suppl 86:8-160. doi: 10.1111/j.1398-9995.2007.01620.x. No abstract available. PMID 18331513